CLINICAL TRIAL: NCT02449460
Title: Multicenter Observational Study of Epidemiology of Cardiovascular Diseases and Risk Factors in Different Regions of Russian Federation
Brief Title: Cardiovascular Epidemiology in Russian Federation
Acronym: ESSE-RF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Collaborators: National Research Center for Preventive Medicine (Other Government); Russian Cardiology Research and Production Center (Other)
Responsible Party: Principal Investigator, Conrady Alexandra, professor, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Other Study IDs: AlmazovFCHBE-4
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Hypertension; Coronary Artery Disease; Diabetes; Heart Failure; Smoking; Lifestyle
Keywords: hypertension; epidemiology; glucose; body mass index; lipids; smoking; coronary artery disease; arterial stiffness; carotid ultrasound
MeSH Terms: conditions — Hypertension; Coronary Artery Disease; Diabetes Mellitus; Heart Failure; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood serum plasma urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study addresses epidemiology of cardiovascular risk factors and major cardiovascular diseases in Russian Federation (urban and rural population). 12 regions of 1600 participants in each will be included.

DETAILED DESCRIPTION:
Plasma lipids and fasting glucose, heart rate and blood pressure, anthropometry, smoking and alcohol questionaries, nutrition, sleep quality, stress will be assessed. ECG records are obtained form all participants. Subclinical target organ damage (carotid and periferal atherosclerosis, pulse wave velocity) will be measured in selected sites. Brain natriuretic peptide, adipose tissue cytokines, hsCRP and genetic markers are also under evaluation

ELIGIBILITY:
Inclusion Criteria:

- informed consent

Exclusion Criteria:

No

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random sample population
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2012-07; Primary Completion 2021-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 10 years
  all cause motality registered by official statistics

SECONDARY OUTCOMES:
Stroke | 10 years
  ischemic and heamorragic stroke
Miocardial infarction | 10 years
Cardiovascular mortality | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana A Shalnova, Prof, Study Chair — State Sientific Center of Preventive Medicine; Alexandra O Konradi, Prof, Principal Investigator — Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health; Eugene I Chazov, Prof, Principal Investigator — Russian Research and Production Complex
Locations (2):
- Russia (2):
  - Orenburg Medical Academi, Orenburg
  - Samara Medical University, Samara